CLINICAL TRIAL: NCT03057691
Title: The Impact of Depression and/or Anxiety on Patients With Acute Coronary Syndrome After Percutaneous Coronary Interventions
Brief Title: The Impact of Depression and/or Anxiety on PCI Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Shaanxi Provincial People's Hospital (Other); The First Hospital of Xi An City (Unknown); Baoji Central Hospital (Other); General Hospital of Ningxia Medical University (Other); The People's Hospital of Ningxia (Other); Wuzhong City People's Hospital (Unknown); LanZhou University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Xinjiang Provincial People's Hospital (Unknown); the First Division Hospital of Xinjiang Production and Construction Corps (Unknown)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF-CRF-2016-004
Record Dates: First submitted 2017-02-15; First posted 2017-02-20 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-10

CONDITIONS: Acute Coronary Syndrome; Depression; Anxiety
Keywords: Acute Coronary Syndrome; Depression; Anxiety; Percutaneous Coronary Intervention; Major Adverse Cardiovascular Events
MeSH Terms: conditions — Acute Coronary Syndrome; Depression; Anxiety Disorders | interventions — Antidepressive Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- No depression/anxiety: patients suffered from ACS who have undergone PCI without depression or anxiety
- Depression: patients suffered from post-ACS depression who have undergone PCI
  Interventions: Other: antidepressive and anti-anxiety therapy
- Anxiety: patients suffered from post-ACS anxiety who have undergone PCI
  Interventions: Other: antidepressive and anti-anxiety therapy
- Depression with anxiety: patients suffered from post-ACS depression with anxiety who have undergone PCI
  Interventions: Other: antidepressive and anti-anxiety therapy

INTERVENTIONS:
Other: antidepressive and anti-anxiety therapy — These therapies include antidepressants, antianxiety drugs and psychotherapy. Subjects choose the therapy follow their own will. All of the above-mentioned therapies are identified by experienced psychiatrists in the same center. The treatment information will be recorded in each visit. The study is considered non-interventional, and no antidepressive or anti-anxiety therapies are mandated.
  Groups: Anxiety; Depression; Depression with anxiety

SUMMARY:
The purpose of this study is to evaluate how depression and/or anxiety could effect the prognosis of the patients post-ACS after PCI.

DETAILED DESCRIPTION:
This trial is a prospective, multi-centric, real-world clinical study. About 5,000 patients with ACS post-PCI will be recruited according to the resource available of each participating center to represent real-world setting. Patients enrolled in the project will accept two-years' follow-up and will be assessed on mortality, cardiovascular events, and severity of depressive or anxiety symptoms using self-rating scales continuously during the trial, in which their treatment for anxiety or depression will also be documented.

ELIGIBILITY:
Inclusion criteria

1. Aged > 18 years old 2. Patients with a diagnosis of ACS including acute myocardial infarction (MI) and unstable angina (UA). Acute MI diagnosis must be met with at least two of these following criteria: typical chest pain, abnormal elevation of cardiac biomarkers, and electrocardiographic changes consist with MI. The diagnosis of UA includes new onset angina within 1 month, crescendo angina, resting angina, infarction angina, and variant angina.

3. Good recovery from PCI. 4. Volunteer for the study and sign the informed consent. Exclusion Criteria

1. Severe heart failure, defined as left ventricular ejection fraction (LVEF)≤30% or New York Heart Association (NYHA) class≥III.
2. Severe renal dysfunction, defined as creatinine clearance rate ≤30 ml/min.
3. Cancer.
4. Other severe mental illness including schizophrenia, severe dementia, substance abuse, etc.
5. Bipolar disorder.
6. Ongoing administration of antipsychotic, antidepressant, or antianxiety drugs.
7. Serious risk of suicide.
8. Severe, life-threatening medical condition (patients cannot participate in the study course).
9. Pregnancy and lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients suffered from acute coronary syndrome after percutaneous coronary intervention
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2017-03-11 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events | From date of first visit until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  death, myocardial infarction, stroke, angina pectoris, revascularization.

SECONDARY OUTCOMES:
Depression self-rating scales | From date of first visit until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  results of depression scales assessed by The Patient Health Questionnaire-2 (PHQ-2, scores ≤2 non, >2 continue PHQ-9) or PHQ-9 (scores ≤4 non, 5~9 mild, 10~19 mediate, ≥ 20 severe)
Anxiety self-rating scales | From date of first visit until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  results of anxiety scales assessed by Generalized Anxiety Disorder 2-item(GAD-2, scores ≤2 non, >2 continue GAD-7) or GAD-7 (scores ≤4 non, 5~9 mild, 10~14 mediate, ≥15 severe)

CONTACTS AND LOCATIONS:
Overall Officials: Zuyi Yuan, Professor, Study Director — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Teply RM, Packard KA, White ND, Hilleman DE, DiNicolantonio JJ. Treatment of Depression in Patients with Concomitant Cardiac Disease. Prog Cardiovasc Dis. 2016 Mar-Apr;58(5):514-28. doi: 10.1016/j.pcad.2015.11.003. Epub 2015 Nov 10. PMID 26562328
- [Background] Lichtman JH, Froelicher ES, Blumenthal JA, Carney RM, Doering LV, Frasure-Smith N, Freedland KE, Jaffe AS, Leifheit-Limson EC, Sheps DS, Vaccarino V, Wulsin L; American Heart Association Statistics Committee of the Council on Epidemiology and Prevention and the Council on Cardiovascular and Stroke Nursing. Depression as a risk factor for poor prognosis among patients with acute coronary syndrome: systematic review and recommendations: a scientific statement from the American Heart Association. Circulation. 2014 Mar 25;129(12):1350-69. doi: 10.1161/CIR.0000000000000019. Epub 2014 Feb 24. PMID 24566200
- [Background] Oldroyd JC, Cyril S, Wijayatilaka BS, O'Neil A, McKenzie DP, Zavarsek S, Sanderson K, Hare DL, Fisher AJ, Forbes AB, Barr Taylor C, Clarke DM, Meredith IT, Oldenburg B. Evaluating the impact of depression, anxiety & autonomic function on health related quality of life, vocational functioning and health care utilisation in acute coronary syndrome patients: the ADVENT study protocol. BMC Cardiovasc Disord. 2013 Nov 17;13:103. doi: 10.1186/1471-2261-13-103. PMID 24237848
- [Background] Regan KL. Depression treatment with selective serotonin reuptake inhibitors for the postacute coronary syndrome population: a literature review. J Cardiovasc Nurs. 2008 Nov-Dec;23(6):489-96. doi: 10.1097/01.JCN.0000338929.89210.af. PMID 18953212
- [Background] Ossola P, Paglia F, Pelosi A, De Panfilis C, Conte G, Tonna M, Ardissino D, Marchesi C. Risk factors for incident depression in patients at first acute coronary syndrome. Psychiatry Res. 2015 Aug 30;228(3):448-53. doi: 10.1016/j.psychres.2015.05.063. Epub 2015 Jun 27. PMID 26144582
- [Background] Huffman JC, Celano CM, Januzzi JL. The relationship between depression, anxiety, and cardiovascular outcomes in patients with acute coronary syndromes. Neuropsychiatr Dis Treat. 2010 May 6;6:123-36. doi: 10.2147/ndt.s6880. PMID 20505844
- [Background] Celano CM, Millstein RA, Bedoya CA, Healy BC, Roest AM, Huffman JC. Association between anxiety and mortality in patients with coronary artery disease: A meta-analysis. Am Heart J. 2015 Dec;170(6):1105-15. doi: 10.1016/j.ahj.2015.09.013. Epub 2015 Sep 21. PMID 26678632
- [Background] Nezafati MH, Vojdanparast M, Nezafati P. Antidepressants and cardiovascular adverse events: A narrative review. ARYA Atheroscler. 2015 Sep;11(5):295-304. PMID 26715935
- [Background] Marke V, Bennett P. Predicting negative emotional states following first onset acute coronary syndrome. J Health Psychol. 2017 May;22(6):765-775. doi: 10.1177/1359105315614996. Epub 2015 Nov 26. PMID 26613707
- [Derived] Xiao Y, Li W, Zhou J, Zheng J, Cai X, Guo M, Hao X, Zhang Z, Liu Y, Yuan Z. Impact of depression and/or anxiety on patients with percutaneous coronary interventions after acute coronary syndrome: a protocol for a real-world prospective cohort study. BMJ Open. 2019 Sep 5;9(9):e027964. doi: 10.1136/bmjopen-2018-027964. PMID 31492778